CLINICAL TRIAL: NCT04965012
Title: Testing the Efficacy of an Online Evidence-Based Treatment for Heavy Cannabis Use in Canadian Adults: A Randomized Controlled Trial (RCT)
Brief Title: Testing the Efficacy of an Online Treatment Program for Heavy Cannabis Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: York University (Other)
Collaborators: University of Manitoba (Other)
Responsible Party: Principal Investigator, Matthew Keough, Assistant Professor, York University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YM8974384y57393848938nv8493478
Record Dates: First submitted 2021-07-06; First posted 2021-07-16 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Marijuana Use; Marijuana Dependence
Keywords: Cannabis; CANreduce; Marijuana; Cognitive Behavioural Therapy; Motivational Enhancement Therapy; Online treatment; Randomized Controlled Trial
MeSH Terms: conditions — Marijuana Use; Marijuana Abuse

STUDY DESIGN:
Intervention Model Description: A three-arm RCT will be conducted to evaluate the proposed online intervention. Eligible participants will be randomized to the CBT with MET condition, the CBT without MET condition, or the psychoeducational control (i.e., control) condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBT with MET treatment group (Experimental): Participants in this arm will be provided with an MET-therapist guided introduction, in addition to the online CBT treatment.
  Interventions: Behavioral: Online CBT with MET treatment
- CBT without MET treatment group (Experimental): Participants in this arm will be provided with a brief non-MET research assistant-led welcome to the program, in addition to the online CBT treatment.
  Interventions: Behavioral: CBT without MET treatment
- Psychoeducation (Control) (No Intervention): The control group will be provided with psychoeducational resources about cannabis and wellbeing.

INTERVENTIONS:
Behavioral: Online CBT with MET treatment — The CBT with MET treatment condition will begin with an MET-therapist guided introduction to the program and first module. After this guided introduction, they will have access to the remaining 7 treatment modules and have 6 weeks to complete them. The content of all modules is derived from Cognitive Behavioural Therapy and Motivational Interviewing. Through module engagement, participants will identify goals related to cannabis use, learn strategies to cope with cravings, triggers, and social pressures, and learn to how prevent relapse. Participants will work through modules sequentially.
  Arms: CBT with MET treatment group
Behavioral: CBT without MET treatment — The CBT without MET treatment condition will begin with a brief non-MET trained research assistant welcome to the program, and will not include working through the first module together. After this welcome, they will have access to the 8 treatment modules and have 6 weeks to complete them. The content of all modules is derived from Cognitive Behavioural Therapy and Motivational Interviewing. Through module engagement, participants will identify goals related to cannabis use, learn strategies to cope with cravings, triggers, and social pressures, and learn to how prevent relapse. Participants will work through modules sequentially.
  Arms: CBT without MET treatment group

SUMMARY:
Cannabis is a frequently-used psychoactive substance. While the majority of individuals can use cannabis without experiencing problems, a small minority of people develop cannabis problems. Despite the small-to-medium reported effect sizes of cognitive behavioural therapy (CBT) and motivational enhancement therapy (MET) treatments for cannabis misuse, many cannabis users do not seek treatment. Online CBT/MET programs have the potential to be cost-effective and accessible, and offer a less stigmatizing option for treatment. These programs may also help capture cannabis users who experience subclinical problems, who are not captured by traditional treatment. Existing treatment programs also need to be adapted to maximize participant retention and increase treatment completion, as many current cannabis use treatment programs have significant drop-out rates. Hence, the goal of the proposed randomized controlled trial (RCT) is to examine the efficacy of an online evidence-based CBT/MET treatment program. Outcomes of a combined CBT/MET treatment program will be compared to a CBT-only treatment program and a waitlist control. This research will provide insight into the novel contribution of MET to online CBT treatment programs for cannabis misuse.

The researchers are hoping to recruit 303 participants for this study from Central and Eastern Canada. Participants will be randomly assigned to one of the treatment groups (i.e., CBT with MET, CBT without MET) or the psychoeducational control group. Individuals in either treatment group will be given 6 weeks to work through 8 online modules. Throughout the modules, participants will identify goals related to cannabis use, learn strategies to cope with cannabis cravings, triggers, and social pressures and learn to prevent relapse. Participants randomly assigned to the control (i.e., psychoeducation) will receive links to websites that provide general psychoeducation about cannabis use and wellbeing. All participants will complete online assessment measures at baseline, end of treatment, and at follow up approximately one month later (i.e., 0 weeks, 6 weeks, 10 weeks) in order to assess the efficacy of the treatment. At the end of the study, individuals in the control group will be given access to the CBT without MET treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ages 19+
* Living in Manitoba or Ontario, Canada
* Reporting moderate difficulties with cannabis as indicated by a score of 8 or more on the Cannabis Use Disorders Identification Test - Revised (CUDIT-R; Adamson et al., 2010)
* Fluency in English
* Having weekly Internet access with a device that allows for video connection
* Self-report at least a 6 out of 10 on a Likert-type scale for motivation to reduce cannabis use (i.e., how important it is to reduce cannabis use)

Exclusion Criteria:

* Self-reported engagement in other psychological or pharmacological treatments for cannabis use
* Elevated suicidality, as defined by scoring greater than minimal risk on a screener
* Current serious psychiatric disorders or history of psychosis, schizophrenia, bipolar disorder
* Are a woman who is currently pregnant or breastfeeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Cannabis Use | Participants will be assessed using the DFAQ-CU at three time points (i.e., prior to treatment; T0); immediately following the 6-week treatment (T1), and at follow-up (i.e., 10 weeks from baseline, 4 weeks from end of treatment, T2).
  The Daily Sessions, Frequency, Age of Onset, and Quantity of Cannabis Use Inventory (DFAQ-CU; Cuttler & Spradlin, 2017) is a self-report inventory of cannabis use that will be used as the primary assessment of cannabis use. The frequency (i.e., number of days per week) and quantity (i.e., grams) of cannabis use subscales will be used. There is mixed evidence as to whether frequency or quantity better predicts cannabis-related severity, thus information on both will be analyzed.

SECONDARY OUTCOMES:
Cannabis-Related Problems | Participants will be assessed using the CUDIT-R at three time points (i.e., prior to treatment; T0); immediately following the 6-week treatment (T1), and at follow-up (i.e., 10 weeks from baseline, 4 weeks from end of treatment, T2).
  The Cannabis Use Disorders Identification Test-Revised (CUDIT-R; Adamson et al., 2010), is an 8-item self-report questionnaire that will be used to assess problematic cannabis misuse characteristic of Cannabis Use Disorder (CUD).
Anxiety | Participants will be assessed using the GAD-7 at three time points (i.e., prior to treatment; T0); immediately following the 6-week treatment (T1), and at follow-up (i.e., 10 weeks from baseline, 4 weeks from end of treatment, T2).
  The General Anxiety Disorder Scale (GAD-7; Spitzer et al., 2006) is a 7-item self-report anxiety questionnaire that will be used to assess overall anxiety severity.
Depression | Participants will be assessed using the PHQ-9 at three time points (i.e., prior to treatment; T0); immediately following the 6-week treatment (T1), and at follow-up (i.e., 10 weeks from baseline, 4 weeks from end of treatment, T2).
  The Patient Health Questionnaire (PHQ-9; Kroenke et al., 2001) is a 9-item self-report of depression symptoms that will be used to assess overall depression severity.
Quality of Life | Participants will be assessed using the WHOQOL-BREF at three time points (i.e., prior to treatment; T0); immediately following the 6-week treatment (T1), and at follow-up (i.e., 10 weeks from baseline, 4 weeks from end of treatment, T2).
  The World Health Organization Quality of Life Assessment (WHOQOL-BREF; WHOQOL Group, 1998) is a 26-item self-report measure that will be used to assess quality of life.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - University of Manitoba, Winnipeg, Manitoba
  - York University, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rysen KK, Carusone JM, Wardell JD, Schaub MP, Wenger A, Wallbridge H, Edgerton JD, Kruk R, Mackenzie CS, Keough MT. Evidence-based therapist guided introduction to online heavy cannabis use treatment in Canadian adults: a Randomized Controlled Trial (RCT). J Cannabis Res. 2026 Jan 17. doi: 10.1186/s42238-025-00378-5. Online ahead of print. PMID 41547862